CLINICAL TRIAL: NCT00743847
Title: A Phase 2 6-Week, Double-Blind, Placebo-Controlled, Multicenter Trial Of Varenicline Tartrate (CP-526,555) For Cognitive Impairment In Subjects With Schizophrenia
Brief Title: A 6-Week Multicenter Trial Of Varenicline Tartrate For Cognitive Impairment In Subjects With Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3051100
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia, treatment, cognition
MeSH Terms: conditions — Schizophrenia | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- varenicline 0.5 mg BID (Active Comparator)
  Interventions: Drug: varenicline
- varenicline 1mg BID (Active Comparator)
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: placebo — Subjects randomized to placebo will receive matching placebo and follow the titration schedule and dosing schedule of those randomized to varenicline.
  Arms: placebo
Drug: varenicline — Subjects randomized to the 0.5 mg arm will be titrated to the full dose during the first week in the following manner: 0.5mg QD x 7 days, then 0.5mg BID for the remainder of the 6 week trial.
  Other Names: Chantix
  Arms: varenicline 0.5 mg BID
Drug: varenicline — Subjects randomized to the 1mg arm will be titrated to the full dose during the first week in the following manner: 0.5mg QD x 3 days, 0.5mg BID x 4 days, then 1mg BID for the remainder of the 6 week trial.
  Other Names: Chantix, Champix
  Arms: varenicline 1mg BID

SUMMARY:
The primary objective of this protocol is to assess the efficacy of two dose strengths of varenicline (0.5 mg BID and 1mg BID) as adjunctive treatment for cognitive impairment in symptomatically stable outpatient schizophrenic subjects who are receiving treatment with atypical antipsychotic medications.

A secondary objective is to evaluate the safety and tolerability of two doses of varenicline in symptomatically stable schizophrenic subjects who are receiving treatment with atypical antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of schizophrenia
* Subjects must be on ongoing maintenance antipsychotic monotherapy or combination therapy with risperidone, olanzapine, quetiapine, ziprasidone, aripiprazole, or paliperidone.
* Evidence of stable symptomatology ≥3 months (eg, no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of symptoms of schizophrenia).

Exclusion Criteria:

* Subjects with a current DSM-IV axis I diagnosis other than schizophrenia.
* Current treatment with conventional antipsychotics (e.g. fluphenazine, haloperidol) or clozapine, or the use of adjunctive anticholinergic treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
CNS Vital Signs Cognition Battery (CNS-VS-M) normed composite score | screening, wk -1, baseline, wk 1,3,6

SECONDARY OUTCOMES:
CNS-VS-M un-normed composite score | screening, wk-1,baseline,wk1,3,6
CNS-VS-M un-normed and normed domain scores | screening, wk-1,baseline, wk1,3,6
University of California San Diego Performance Skills Assessment Brief (UPSA-B) total score | baseline, wk 1,3,6
Severity Item for Cognitive Impairment-Clinician and Patient Versions (SICI-CV; SICI-PV) | baseline, wk6
Global Improvement in Cognition Clinician and Patient Versions (GIC-CV;GIC-PV) | wk 1,3,6
Safety assessments, including adverse events, electrocardiographic assessments, neuropsychiatric assessments (performed weekly), physical exam, and laboratory measures | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051100&StudyName=A%206-Week%20Multicenter%20Trial%20Of%20Varenicline%20Tartrate%20For%20Cognitive%20Impairment%20In%20Subjects%20With%20Schizophrenia